CLINICAL TRIAL: NCT06146309
Title: Assessment Of Peri-papillary Retinal Nerve Fiber Layer Thickness In Patients With Unilateral Branch Retinal Vein Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Akram Fekry Elgazzar, Principal Investigator, Al-Azhar University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Unilateral Branch Retinal Vein
Record Dates: First submitted 2023-11-18; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Branch Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with unilateral BRVO (Experimental)
  Interventions: Drug: aflibercept (2mg/0.05ml)
- Healthy individuals (No Intervention)

INTERVENTIONS:
Drug: aflibercept (2mg/0.05ml) — Aflibercept is a medication used to treat and manage neovascular age-related macular degeneration, diabetic macular edema, myopic choroidal neovascularization, macular edema associated with retinal vein occlusion, and diabetic retinopathy. It is in the vascular endothelial growth factor-A (VEGF-A) and placental growth factor (PlGF) antagonist class of medications. Aflibercept acts as a soluble protein decoy for VEGF receptors to inhibit the predominant signaling pathway responsible for angiogenesis and vascular leakage. Aflibercept and other anti-VEGF inhibitors have become the gold standard in controlling neovascular (wet) age-related macular degeneration (NVAMD). T
  Arms: Patients with unilateral BRVO

SUMMARY:
Several studies have indicated a relation between the development of RVO and elevated intraocular pressure (IOP) and glaucoma [9]. Further investigations into the structural alterations in the fellow eyes of individuals with unilateral RVO have revealed that the pRNFL is thinner than in healthy eyes, suggesting that there may be systemic risk factors for both RVO and glaucoma

ELIGIBILITY:
Inclusion Criteria:

* patients with unilateral BRVO

Exclusion Criteria:

* History of retinal and/or optic nerve diseases involving glaucomatous optic disc, ischemic optic neuropathy, or optic neuritis.
* History of trauma, intravitreal injections, vitreoretinal surgeries, and retinal or macular lasers.
* A significant media opacity that makes it difficult to capture clear images.
* No history of diabetes and/or hypertension in those recruited as the control group

Ages: 47 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
peri-papillary retinal nerve fiber layer thickness | Base line
  Layer of the retina. The thickness was measured by Optical Coherence Tomography
peri-papillary retinal nerve fiber layer thickness | 6 months post injection
  Layer of the retina. The thickness was measured by Optical Coherence Tomography
peri-papillary retinal nerve fiber layer thickness | 12 months post injection
  Layer of the retina. The thickness was measured by Optical Coherence Tomography
peri-papillary retinal nerve fiber layer thickness | 24 months post injection
  Layer of the retina. The thickness was measured by Optical Coherence Tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Akram Fekry Elgazzar, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided